CLINICAL TRIAL: NCT02434705
Title: Protocol for Food Antigen Staining in Esophageal Mucosa in Patients With Eosinophilic Esophagitis
Brief Title: Food Antigen in Eosinophilic Esophagitis
Acronym: EoE
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Joseph A. Murray, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 15-000883
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Antigens

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Antigen (wheat base soy sauce) spray: 1. Ten patients with active and ten with inactive eosinophilic esophagitis (defined by consensus guidelines) undergoing clinically indicated endoscopy and esophageal biopsies will participate in this study.
  2. During the endoscopy two biopsies will be taken from the esophageal body, 10 cm above the gastroesophageal junction.
  3. After biopsies are taken, approximately 10 cc of wheat based soy sauce (antigen spray) will be sprayed though an endoscopic catheter onto the esophageal mucosa. The endoscopic examination will be completed and two additional endoscopic biopsies will be taken 10 cm above the gastroesophageal junction.
  Interventions: Other: Antigen (wheat base soy sauce) spray

INTERVENTIONS:
Other: Antigen (wheat base soy sauce) spray — Patients having a clinically indicated endoscopy for Eosinphilic Esophagitis will have two biopsies from the esophageal body, 10 cm above the gastroesophageal junction. After biopsies are taken, approximately 10 cc of wheat based soy sauce will be sprayed though an endoscopic catheter onto the esophageal mucosa. The endoscopic examination will be completed and Two additional endoscopic biopsies will be taken 10 cm above the gastroesophageal junction.
  Other Names: Wheat based soy sauce

SUMMARY:
The relationship or effect of food antigen (wheat based soy sauce) in eosinophilic esophagitis. It is believed that when food antigens are exposed to the esophageal tissue it starts an chronic allergy-based inflammation. This will be analyzed with the esophageal biopsies and the mucosal impedance probe.

DETAILED DESCRIPTION:
One of the putative mechanisms of eosinophilic esophagitis is exposure of food antigens to antigen recognition cells in the esophageal mucosa that initiates a chronic allergy-based inflammatory response . It is believed that this exposure is facilitated through dilation of the intercellular spaces (DIS) between esophageal epithelial cells (termed spongiosis). This is substantiated by several studies which have demonstrated that: first, DIS is commonly found in biopsies from patients with active EoE and reverses with steroid therapy; second, DIS correlates to physiologic demonstration of increased esophageal epithelial permeability as shown through transepithelial small molecule flux in mucosal biopsies appraised in Ussing chambers and increased conductivity of electric current as measured in a mucosal impedance probe (Katzka, et al., in press, Clin Gastroenterol Hepatol). Although these mechanisms make intuitive sense, no one has shown the presence of food antigen in esophageal mucosa after ingestion and the correlation of this presence to dilation of intercellular spaces.

ELIGIBILITY:
Inclusion criteria:

* Patients between the ages of 18 and 80 with eosinophilic esophagitis diagnosed by a combination of compatible symptoms, endoscopic findings, histology, and lack of response to proton pump inhibitors.
* Patients previously diagnosed with Eosinophilic Esophagitis and are now in histologic remission due to treatment and have <15 eos hpf.

Exclusion Criteria

* Acute allergy to wheat or soy
* Currently taking steroids
* Inability to read due to: Blindness, cognitive dysfunction, or English language illiteracy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eosinophilic Esophagitis patients
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Measurement of Gluten and Soy Antigen in Esophageal Mucosa | one year
  Cryosectioning of the frozen esophageal tissue will then be done for immunofluorescent staining to determine the distribution/localization of different cells and dietary proteins We will use anti-gliadin (Biorbyt catalog # orb157160)and anti-soy (LifeSpan Biosciences Catalog # LS-C132165-100)antibodies against cell surface markers as well as dietary proteins/peptides tagged with different fluorochromes to achieve this.

SECONDARY OUTCOMES:
Dilated intercellular spaces (spongiosis) | one year
  Is graded on the basis of the worst area, using a 0-4+ scale [3]. DIS grading was assessed by the appearance of the tight junctions seen on biopsy and the degree of widening between epithelial cells . Grade 0: no intercellular space widening and intact tight junctions. Grade 1: mild widening of intercellular spaces with attenuation and prominence of tight junctions. Grade 2: Further widening of intercellular space with some disruption of tight junctions. Grade 3: complete disruption of tight junctions with further widening of intercellular spaces, forming small "lakes" in the epithelium. Grade 4: Coalescence of epithelial lakes.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Murray, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials